CLINICAL TRIAL: NCT05328362
Title: CanCope: Digital Intervention for Coping With Cannabis Craving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00032248
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-09

CONDITIONS: Cannabis Use

STUDY DESIGN:
Intervention Model Description: Micro-Randomized Trial (MRT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CanCope Intervention (Experimental): The CanCope intervention was delivered through the MetricWire app which was available to each participant on their personal smartphone. The intervention included a "push" component which was responsive to a participant's level of craving (based on self-report assessed via EMA) and sent messages to each participant via the MetricWire app according to a decision rule. MetricWire randomized delivery of the push component with a probability of 0.33 for receiving a mindfulness coping strategy, 0.33 for receiving a distraction coping strategy, and 0.33 for receiving a thank-you message (attention control) at each decision point when participants were available for the intervention.
  Interventions: Behavioral: CanCope

INTERVENTIONS:
Behavioral: CanCope — Messages prompted participants to use mindfulness-based or distraction-based coping strategies, or a thank-you message which served as an attention control. If participants reported elevated craving (4 or greater) prior to a decision point, they received either a coping strategy message or a control message. If participants reported craving levels of less than 4 they received a control message.

SUMMARY:
The CanCope Study is a micro-randomized trial conducted to gather evidence about and compare the effectiveness of a momentary intervention to help young adults cope with cannabis cravings as they attempt to reduce their use.

DETAILED DESCRIPTION:
The CanCope Study is designed to test the effectiveness of two distinct strategies (mindfulness and distraction) to cope with cannabis cravings in young adults (19 - 25 years) who are attempting to reduce their cannabis use. Cannabis use is determined using a single-item question about the number of days out of the past 30 days the individual used cannabis. Young adults who reported using cannabis >10 out of the past 30 days, who were not pregnant or breastfeeding, and who were not currently in treatment for problems related to substance use were eligible to enroll in this four-week study.

The CanCope intervention was delivered to participants through the MetricWire app, which was available for download on the participants' personal smartphones. Participants were asked to complete five ecological momentary assessments (EMA) per day, which asked questions related to cannabis use including one question about current level of craving on a scale of 0 - 10. If a participant reported a craving level >4, a message was sent via the app encouraging the participant to try a mindfulness or distraction coping strategy, or the participant received a thank-you for completing the EMA which served as an attention control.

ELIGIBILITY:
Inclusion Criteria:

* Used cannabis at least 10 out of the past 30 days

Exclusion Criteria:

* Currently pregnant or breastfeeding
* Currently in treatment for problems related to substance use

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Stanger, PhD, Study Director — Dartmouth College
Locations (1):
- Center for Technology and Behavioral Health, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stanger C, Anderson MAB, Xie H, Nnaka T, Budney AJ, Qian T, Yap JRT, Nahum-Shani I. Momentary mindfulness versus distraction coping messages to reduce cannabis craving among young adults: A microrandomized trial. Psychol Addict Behav. 2025 Mar;39(2):200-211. doi: 10.1037/adb0001029. Epub 2024 Oct 17. PMID 39418443

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants consented to the study in the app prior to completing any eligibility screening measures. Participants who consented but then failed to complete screening or any EMA assessments were not enrolled. EMA completion was required to randomize individual decision points (completed EMAs) to an intervention in this study design. N=53 were enrolled based on these criteria.
Period: Overall Study
Arm/Group | CanCope Intervention
Started | 53
Completed | 49
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Participants who consented in the app but then failed to complete screening/baseline measures or any EMA assessments were not enrolled. EMA completion was required to randomize individual decision points (completed EMAs) to an intervention in this study design. N= 53 were enrolled based on these criteria.
Arm/Group | CanCope Intervention
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.04 (1.97)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Man | 27
  Gender: Woman | 20
  Gender: Nonbinary | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 42
  More than one race | 5
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Average Craving Level - Active vs. Control Messages
Description: Participants were asked to rate their level of cannabis craving on a scale of 0 - 10 five times per day where higher scores indicate more craving. Participants were considered available for randomization when craving >=4 and they clicked the intervention message in the study app. To determine the effect of messaging on craving, we will calculate the average craving level for each EMA eligible for intervention and randomized to receive an active coping strategy message or a control message. It was pre-specified based on a priori power analyses for this small pilot study to combine the "mindfulness-based coping strategies" and "distraction-based coping strategies" interventions in the "Active Message" Row". Craving levels will be averaged across randomized observations. There were up to 140 decision points (5 EMAs per day x 28 days) per participant for the intervention period.
Time Frame: Minimum 2.8 hours after each decision point; Maximum 12.8 hours after each decision point
Population: Only participants who completed baseline measures and at least one ecological momentary assessment (EMA) are included in the analyses. Two participants who completed baseline measures did not complete any EMAs which were required for micro-randomization and are therefore not included in the analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CanCope Intervention: The CanCope intervention was delivered through the MetricWire app which was available to each participant on their personal smartphone. The intervention included a "push" component which was responsive to a participant's level of craving (based on self-report assessed via EMA) and sent messages to each participant via the MetricWire app according to a decision rule. MetricWire randomized delivery of the push component with a probability of 0.67 for receiving an active message (either a mindfulness or a distraction coping strategy), and 0.33 for receiving a thank-you message (attention control) at each decision point when participants were available for the intervention.
  CanCope: Active Messages prompted participants to use mindfulness-based or distraction-based coping strategies, or a thank-you message which served as an attention control. If participants reported elevated craving (4 or greater) and clicked the intervention message, they received either an active coping strategy message or a control message. If participants reported craving levels of less than 4 they received a control message. It was pre-specified to combine the "mindfulness-based coping strategies" and "distraction-based coping strategies" interventions in the "Active Message" category for primary analyses. The study was powered a priori to detect differences in active vs. control messages.
Arm/Group | CanCope Intervention
Number analyzed (Participants) | 53
score on a scale
  Control Message | 4.736 (2.822)
  Active Message | 4.629 (2.780)

ADVERSE EVENTS:
Time Frame: Duration of the study (28 days)
Description: Data about adverse events collected non-systematically (participant report).
Arm/Group | CanCope Intervention
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT05328362/Prot_SAP_000.pdf